CLINICAL TRIAL: NCT02854475
Title: Confocal Raman Spectroscopy: in Vivo Measurement of Physiological Skin Parameters - A Pilot Study
Brief Title: Confocal Raman Spectroscopy: in Vivo Measurement of Physiological Skin Parameters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vienna (Other)
Collaborators: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Lisa Binder, Mag. pharm., University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: Raman 2016.1
Record Dates: First submitted 2016-07-27; First posted 2016-08-03 (Estimated); Last update posted 2016-08-03 (Estimated); Status verified 2016-07

CONDITIONS: Dermatologic Disorders; Disorder of Cholesterol Metabolism
Keywords: skin parameters; cholesterol; Raman spectroscopy
MeSH Terms: conditions — Skin Diseases | interventions — Spectrum Analysis, Raman

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Proband group (Experimental): Raman spectroscopy and venous blood collection
  Interventions: Procedure: Venous blood collection; Procedure: Raman spectroscopy

INTERVENTIONS:
Procedure: Venous blood collection — weekly within two weeks
Procedure: Raman spectroscopy — weekly within two weeks, on the volar forearm, using a RiverDiagnostics gen2-SCA Skin Composition Analyzer

SUMMARY:
The purpose of this study is to

I. determine several skin parameters, for example natural moisturizing factor (NMF) and cholesterol, with Raman spectroscopy in vivo and

II. compare the results with the corresponding cholesterol levels measured in venous blood.

DETAILED DESCRIPTION:
In vivo Raman experiments will be carried out weekly on voluntary participants using a RiverDiagnostics gen2-SCA Skin Composition Analyzer (RiverDiagnostics, Rotterdam, Netherlands). All experiments will be carried out on the volar forearm. Semi-quantitative concentration profiles for several skin parameters will be determined, for example natural moisturizing factor (NMF) and cholesterol.

Additionally the total cholesterol level will be detected by venous blood sample analysis. The blood samples will be taken weekly within two weeks, similar to the Raman measurements.

ELIGIBILITY:
Inclusion Criteria:

* Provision of subject informed consent
* Female or male aged between 18 and 65 years

Exclusion Criteria:

* Pregnancy
* Chronic skin conditions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-07; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Correlation of the fasting total cholesterol levels measured in skin with confocal Raman spectroscopy and in venous blood collected by venipuncture | 2 weeks

SECONDARY OUTCOMES:
Concentration curves of various skin substances, such as NMF, urea and water as evidence for the eligibility of confocal Raman spectroscopy for the in vivo measurement of skin | 2 weeks

IPD SHARING:
Plan to Share IPD: Undecided